Official title: Evaluation of the clinical and molecular efficacy of daily avanafil in Egyptian males with erectile and endothelial dysfunction (Randomized Placebo-Controlled study)

NCT number: NCT04374994

**Document date: 20-9-2018** 

Statistical analysis of the data: Data were fed to the computer and analyzed using IBM SPSS software package version 20.0. Qualitative data were described using number and percent. Quantitative data were described using range (minimum and maximum), mean, standard deviation and median. Significance of the obtained results was judged at the 5% level. Student t-test was used for normally distributed quantitative variables, to compare between two studied groups. Mann Whitney test for abnormally distributed quantitative variables, to compare between two studied groups. Wilcoxon signed ranks test, for abnormally distributed quantitative variables, to compare between two periods. Paired t-test for normally quantitative variables, to compare between two periods Spearman coefficient for correlation between two abnormally quantitative variables.